CLINICAL TRIAL: NCT01312662
Title: Towards Worldwide Comparability of Visual Acuity Assessment A Pilot Study Comparing ETDRS Visual Acuity Charts, Projected Landolt Charts and the Freiburg Visual Acuity Test (FrACT) With a View to Developing a Mathematical Transformation Routine Between the Results From These Three Tests
Brief Title: Towards Worldwide Comparability of Visual Acuity Assessment
Acronym: VisComp
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University of Freiburg (Other)
Responsible Party: Prof. Dr. med. Schiefer, Institute for Ophthalmic Research, University of Tübingen
Other Study IDs: VisComp01
Record Dates: First submitted 2011-03-08; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Comparison of Visual Acuity Tests.; ETDRS. FrACT. Landolt Rings.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- normal ophthalmological status
- opacity of the refractive media
- maculopathy
- optic neuropathy
- chiasmal and postchiasmal visual pathway pathologies
- amblyopia (deprivation)
- amblyopia (strabism)

SUMMARY:
Purpose of this study is to investigate the agreement, the test-retest reliability of three established and widely used visual acuity tests, to develop a mathematical transformation routine between the results from these three tests, to assess the examinees´ and examiners´ acceptance and to compare the test durations.

DETAILED DESCRIPTION:
Assessment of distant visual acuity is the most frequently used procedure for estimation of visual performance. However, there exist a vast number of markedly differing visual acuity tests worldwide; furthermore there are differing report formats to express acuity. This variety may critically interfere with standardization and comparability of this basic visual test method.

Purpose of this study is to investigate the agreement, the test-retest reliability of three established and widely used visual acuity tests, i.e., the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts, a conventional projected distant visual acuity test according to DIN 58220 part 3, and the Freiburg visual acuity test (FrACT), to develop a mathematical transformation routine between the results from these three tests, to assess the examinees´ and examiners´ acceptance and to compare the test durations.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of:

* normal ophthalmological status,
* opacity of the refractive media,
* maculopathy,
* optic neuropathy
* chiasmal and postchiasmal visual pathway pathologies,
* amblyopia (deprivation),
* amblyopia (strabism)

Exclusion Criteria:

* underage person
* concomitance of different eye-diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University eye Hospital Tuebingen
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2011-03

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Ophthalmic Research, University of Tuebingen, Tübingen, Germany